CLINICAL TRIAL: NCT04504578
Title: Efficacy and Safety of Contact Lens-assisted Corneal Cross- Linking in the Treatment of Keratoconus With Thin Corneas
Brief Title: Efficacy and Safety ofCACXL in the Treatment of Keratoconus With Thin Corneas
Acronym: CACXL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Moustafa Nour, assistant lecturer, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s5-2019
Record Dates: First submitted 2020-07-05; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Progressive Keratoconus
Keywords: cross linking; thin corneas; Advanced keratoconus

STUDY DESIGN:
Intervention Model Description: patients with progressive keratoconus with thin corneas less than 400 micron
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with progressive keratoconus with thin corneas (Experimental): patients with progressive keratoconus with thin corneas , with thickness less than 400 micron ,will do conventional cross linking but with putting contact lens over the cornea ( will receive Contact lens assisted corneal cross liking )
  Interventions: Procedure: contact lens assisted corneal cross linking

INTERVENTIONS:
Procedure: contact lens assisted corneal cross linking — 40 eyes of 30 patients underwent CACXL. The central 9 mm of corneal epithelium was abraded , Iso-tonic riboflavin 0.1% was applied every 2 minutes for 10 minutes on the debrided cornea. A disposable soft Contact lens without an ultraviolet filter (Soflens, Bausch & Lomb) was placed in the inferior fornix during soaking of the stroma with riboflavin for 10 minutes. The contact lens was applied on the corneal surface and the cornea was exposed to ultraviolet-A irradiation at fluence of 3.0 mW/cm2 for 30 minutes The uncorrected (UDVA) and best corrected (BDVA) visual acuity, and maximum (K max) keratometric values, were assessed before, and after 9 months CXL. Endothelial cell count was assessed before and 3 months after CXL. Anterior segment OCT was done 1 month after CXL to evaluate the presence and depth of the corneal stromal demarcation line.

SUMMARY:
The aim of this study is to detect the safety and effectiveness of contact lens assisted corneal cross linking in managing progressive keratoconus with thin corneas CACXL was done for 40 eyes of 30 of keratoconic patients presented to cornea outpatient clinic in Kasr Alainy teaching hospital The UDVA ,BDVA KMAX, thinnest corneal thickness pre-operative and 9 months postoperatively and the endothelial cell count was measured preoperative and 3 months postoperative Demarcation line was measured after 1 month by using ASOCT There was statistical significant difference in UDVA and BDVA, there was stabilization of Kmax there was decrease in endothelial cell count but not statistically significant According to results the procedure seems to be effective and safe un managing progressive keratoconus.

DETAILED DESCRIPTION:
Corneal collagen cross linking showed effective results in stabilizing progressive keratoconic corneas. It is the only treatment that halts progression of keratoconus, It was first described in 1998 by Spoerl et al . A major limitation of the procedure that it cannot be used in corneas with pachymetry less than400 micrometers based on the fact that an irradiance of 0.37 mW/cm2 has been found to be cytotoxic for the endothelial cell layer. Since the absorption coefficient for the human corneas is 70 cm-1 and the intended surface irradiance is 3.0 mW/cm2, the 0.37 mW/cm2 irradiance is reached at 300 microns depth. In a 400 microns thick cornea saturated with riboflavin, the irradiance at the endothelial level is 0.18 mW/cm2, which is a factor of 2 smaller than the damage threshold. Therefore, the 400 microns limit is considered to be a safe limit to protect the endothelium and intraocular structures from the hazards of UV irradiation 12 However , the patients with advanced ectasia who are desperately in need for cxl , are the same ones who have thin corneas often below the threshold which is considered to be safe for CXL treatment However further studies with longer follow up and larger numbers of cases are needed to confirm our findings.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 35years old Mild , moderate and severe keratoconic patients with a corneal thickness from 360-400 µm at the thinnest location .

Exclusion Criteria:

* • Previous corneal surgeries such as rings or crosslinking.

  * Patients with stromal corneal scar.
  * Other ocular pathology such as glaucoma or iridocyclitis.
  * Patient with systemic diseases that likely affects wound healing such as insulin dependent diabetes mellitus.
  * Patients with collagen vascular diseases, autoimmune or immune deficiency diseases.
  * Pregnant or nursing women.
  * Patients taking the following medications ; isotretinoin, amiodarone, sumatriptan.
  * Other corneal pathology rather than keratoconus

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
kmax | tomography after 9 months
  stabilization of the cornea by corneal tomography

SECONDARY OUTCOMES:
number of endothelial cell count | 3 months postoperative by specular microscopy
  number of endothelial cell before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kasrelaini Hospital, Cairo, Egypt

REFERENCES:
- [Derived] Nour MM, El-Agha MH, Sherif AM, Shousha SM. Efficacy and Safety of Contact Lens-Assisted Corneal Crosslinking in the Treatment of Keratoconus With Thin Corneas. Eye Contact Lens. 2021 Sep 1;47(9):500-504. doi: 10.1097/ICL.0000000000000799. PMID 34001713